CLINICAL TRIAL: NCT06200519
Title: A Longitudinal Observational Assessment of Diastolic Function During the Transitional Period and Infancy Using Serial Echocardiography in Neonates Born at 35 Weeks Gestation or Above
Brief Title: Assessment of Diastolic Function During the Transitional Period and Infancy Using Serial Echocardiography
Acronym: DiFuSE
Status: Not yet recruiting | Type: Observational
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Dr. Gene Dempsey, Horgan Chair in Neonatology, Consultant Neonatologist, University College Cork
Other Study IDs: DiFuSE
Record Dates: First submitted 2023-12-21; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Diastolic Dysfunction; Neonatal Encephalopathy; Small for Gestational Age at Delivery; Transient Tachypnea of the Newborn; Trisomy 21; Gestational Diabetes
Keywords: Diastolic function; Neonatal transition; Longitudinal; Tissue Doppler imaging; Speckle tracking echocardiography
MeSH Terms: conditions — Transient Tachypnea of the Newborn; Down Syndrome; Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neonates born at 35 weeks gestation and above: Stratification of population for recruitment and data analysis
  1. Gestational age in weeks
  2. Birth weight and centile
  3. Small for gestational age (birth weight <10th centile post-natal)
  4. Large for gestational age (birth weight >90th centile post-natal)
  5. Evidence of antenatal Doppler abnormalities
  6. Maternal gestational diabetes mellitus or pre-existing diabetes mellitus
  7. Maternal pre-eclampsia
  8. Signs of maternal chorioamnionitis
  9. Mode of delivery
  10. Transient Tachypnea of Newborn
  11. Pregnancy conceived by assisted reproductive technologies
  12. Maternal medication use
  13. Suspected or confirmed Trisomy 21
  14. Gestational age at birth 35-36+6 gestation group
  15. Feeding type
  16. Mild neonatal encephalopathy
  17. Moderate and severe neonatal encephalopathy receiving therapeutic hypothermia

SUMMARY:
The goal of this single-centre longitudinal observational study is to create reference values for diastolic function parameters in neonates born at 35 weeks' gestation or above, and to assess the influence of pre-defined antenatal, intrapartum, maternal, and neonatal factors on cardiac function.

The main question it aims to answer are:

* What are the normal reference ranges for parameters of diastolic cardiac function in neonates?
* How are these influenced by maternal, intrapartum and neonatal factors?
* Do the diastolic changes noted during the first two days of life persist into infancy?

Participants will have four echocardiographic assessments in total:

* Two during the first 48 hours of life (prior to discharge home)
* Two during infancy (as an outpatient)

DETAILED DESCRIPTION:
Participants will have their first echo to assess diastolic function, using both conventional and novel echocardiographic measure, within the first 6 to 18 hours of life approximately (Day 1 scan) and this will be repeated at 30 to 42 hours of life (Day 2 scan). Both scans will involve a comprehensive structural assessment to confirm normal anatomy.

All participants will be invited to return for follow-up targeted echocardiography assessments to evaluate function at approximately 6 - 9 months (Scan 3) and at approximately 12 - 18 months of life (Scan 4). At each of these visits, their weight, height, any interim hospital admissions, serious illnesses or medical issues and medications will be documented using a structured checklist format.

ELIGIBILITY:
Inclusion Criteria:

* Birth at 35 weeks gestation or above
* Informed consent obtained

Exclusion Criteria:

* Any apparent congenital anomalies
* Any known chromosomal abnormalities (except Trisomy 21)
* Any known congenital structural heart disease (except patent ductus arteriosus, atrial septal defect, patent foramen ovale or ventricular septal defect)

Ages: 6 Hours to 18 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All neonates greater than or equal to 35 weeks gestational age at birth and who meet the inclusion and exclusion criteria in Table 1 below will be considered for inclusion. Informed consent will be obtained from the parent prior to inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Reference values for diastolic function parameters in neonates | Day 1 and Day 2 of life
  Establish reference values for conventional and novel echocardiographic methods of assessing diastolic function in neonates and stratify them by different antenatal, intrapartum, maternal and neonatal factors to assess whether there is an association between these factors and cardiac function.
Persistence of diastolic function changes into infancy | 6 - 9 months of life, 12 - 18 months of life
  Assess whether the diastolic function changes noted in the first few days persist over time.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Dempsey, Principal Investigator — University College Cork
Locations (1):
- Cork University Maternity Hospital, Cork, Ireland

REFERENCES:
- [Background] Breatnach CR, Levy PT, James AT, Franklin O, El-Khuffash A. Novel Echocardiography Methods in the Functional Assessment of the Newborn Heart. Neonatology. 2016;110(4):248-260. doi: 10.1159/000445779. Epub 2016 Jun 10. PMID 27287615
- [Background] Kozak-Barany A, Jokinen E, Rantonen T, Saraste M, Tuominen J, Jalonen J, Valimaki I. Efficiency of left ventricular diastolic function increases in healthy full-term infants during the first months of life. A prospective follow-up study. Early Hum Dev. 2000 Jan;57(1):49-59. doi: 10.1016/s0378-3782(99)00057-2. PMID 10690711
- [Background] Khot N, Joshi S, Malwade S, Chavan S, Mane SV, Agarkhedkar S, Arora A. A Comprehensive Echocardiographic Assessment of Neonatal Right Ventricular Function in Neonatal Intensive Care Unit Babies. Cureus. 2023 Apr 5;15(4):e37166. doi: 10.7759/cureus.37166. eCollection 2023 Apr. PMID 37153277
- [Background] Tao K, Hara Y, Ishihara Y, Ohshima Y. Cesarean section predominantly affects right ventricular diastolic function during the early transitional period. Pediatr Neonatol. 2019 Oct;60(5):523-529. doi: 10.1016/j.pedneo.2019.01.004. Epub 2019 Jan 19. PMID 30713044
- [Background] Verma A, Suryawanshi P, Chetan C, Oka G, Singh Y, Kallimath A, Singh P, Garegrat R. A detailed echocardiographic evaluation of ventricular functions in stable full term small for gestational age babies. J Ultrasound. 2023 Mar;26(1):117-127. doi: 10.1007/s40477-022-00691-2. Epub 2022 May 26. PMID 35616853
- [Background] Sirc J, Dempsey EM, Miletin J. Diastolic ventricular function improves during the first 48-hours-of-life in infants weighting <1250 g. Acta Paediatr. 2015 Jan;104(1):e1-6. doi: 10.1111/apa.12788. Epub 2014 Oct 2. PMID 25163391
- [Background] Vrancken SL, van Heijst AF, de Boode WP. Neonatal Hemodynamics: From Developmental Physiology to Comprehensive Monitoring. Front Pediatr. 2018 Apr 5;6:87. doi: 10.3389/fped.2018.00087. eCollection 2018. PMID 29675404
- [Derived] Stapleton I, Bussmann N, Finn D, Livingstone V, Dempsey E. Assessment of Diastolic Function during the transitional period and infancy using Serial Echocardiography in a tertiary neonatal unit (DiFuSE): a longitudinal prospective observational study protocol. BMJ Open. 2025 Aug 19;15(8):e095984. doi: 10.1136/bmjopen-2024-095984. PMID 40829821